CLINICAL TRIAL: NCT06344455
Title: Influence of Educational Stimuli From the Pé-de-Meia Program on Delay Discounting Propensity: A Study With the Modified Iowa Gambling Task
Brief Title: Influence of Educational Stimuli From the Pé-de-Meia Program on Delay Discounting Propensity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal Institute of Education, Science and Technology of the State of Mato Grosso (Other)
Responsible Party: Principal Investigator, Pamela Rodrigues Miranda, PROFESSOR, Federal Institute of Education, Science and Technology of the State of Mato Grosso
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RCT Delay Discounting
Record Dates: First submitted 2024-03-15; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Delay Discounting

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Convergent Group (Experimental)
  Interventions: Behavioral: School Retention and Completion Incentive Savings via Modified Iowa Gambling Task A
- Divergent Group (Experimental)
  Interventions: Behavioral: School Retention and Completion Incentive Savings via Modified Iowa Gambling Task B
- Control Group (Placebo Comparator)
  Interventions: Behavioral: Iowa Gambling Task

INTERVENTIONS:
Behavioral: School Retention and Completion Incentive Savings via Modified Iowa Gambling Task A — Participants will engage in a modified version of the Iowa Gambling Task with visual stimuli that are aligned with the Pé-de-Meia program's requirements. Advantageous cards will display images that are congruent with the program's criteria, while disadvantageous cards will feature images that are contrary to the Pé-de-Meia program's requirements.
  Arms: Convergent Group
Behavioral: Iowa Gambling Task — The participants will play the unmodified Iowa Gambling Task.
  Arms: Control Group
Behavioral: School Retention and Completion Incentive Savings via Modified Iowa Gambling Task B — The participants will play the modified IGT (Iowa Gambling Task). For the disadvantageous cards, images that align with the requirements of the "Pé-de-Meia" program will be presented, while for the advantageous cards, images that contradict the criteria of the "Pé-de-Meia" program will be shown.
  Arms: Divergent Group

SUMMARY:
The goal of this randomized clinical trial is to investigate how the Stay-and-Complete School Incentive Savings, part of the Pé-de-Meia Program, affects decision-making among low-income high school students, particularly their tendency towards delay discounting. This concept describes the preference for immediate gratifications over larger future rewards. The main questions it seeks to answer are:

Can exposure to the specific educational stimuli of the Pé-de-Meia Program alter students' propensity for delay discounting? How do different levels of delay discounting influence students' decision-making regarding their studies and the utilization of the program's incentives?

Participants will:

Engage in a modified version of the Iowa Gambling Task (IGT), a computerized game that simulates decision-making under uncertainty, adapted to reflect the stimuli and choices related to the Pé-de-Meia Program.

Complete questionnaires that measure their propensity for delay discounting and gather demographic and socioeconomic information.

Researchers will compare the outcomes among groups of students exposed to different types of stimuli (aligned with the program's objectives, contrasting, and a control group without modifications) to see if the specific financial and educational incentives of the Pé-de-Meia Program influence how students value immediate rewards compared to future benefits. This study is expected to contribute to the improvement of public educational policies, encouraging school retention and promoting the educational success of low-income adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Low-income high school students in the public system, registered in CadÚnico

Exclusion Criteria:

* Students with a formal psychological or psychiatric diagnosis

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Delay Discounting 1 | up to 12 weeks
  measured by the Monetary Choice Questionnaire (MCQ). 0.0 indicates an absence of discounting, meaning the individual values immediate and future rewards equally. This can be interpreted as a preference for delayed rewards or a long-term perspective.
  0.5 indicates strong discounting, meaning the individual significantly devalues future rewards in favor of immediate ones. This is seen as an indication of high impulsivity
Delay Discounting 2 | up to 24 weeks
  measured by the Monetary Choice Questionnaire (MCQ). 0.0 indicates an absence of discounting, meaning the individual values immediate and future rewards equally. This can be interpreted as a preference for delayed rewards or a long-term perspective.
  0.5 indicates strong discounting, meaning the individual significantly devalues future rewards in favor of immediate ones. This is seen as an indication of high impulsivity

SECONDARY OUTCOMES:
decision-making performance under risk and uncertainty | up to 24 weeks
  It will be calculated according to the standard scoring approach that evaluates long-term decision-making, considering the number of advantageous choices (deck C + D) minus the number of disadvantageous choices (deck A + B) over 100 trials. The higher the net financial value accumulated over time, the better the performance.
  Therefore, the "best performance" in the IGT can more appropriately be defined as the outcome that provides the greatest net financial return at the end of the choices. This reflects the participant's ability to effectively manage risks and rewards, prioritizing choices that maximize financial gains over time, despite the fluctuations and uncertainties inherent to each choice.
loss aversion | up to 24 weeks
  Loss aversion will be measured through the Iowa Gambling Task, by the proportion of choices that avoid large losses. The minimum value (0) would indicate no loss aversion (i.e., the participant chooses equally among all decks, without avoiding the large losses). The maximum value (1, or 100%) would indicate a complete loss aversion (i.e., the participant always avoids choosing the decks with large potential losses).
  A higher score in this context would indicate a greater aversion to loss, meaning that the participant is more inclined to avoid choices that could result in large losses, even if this may limit their potential gains.
Loss Frequency-Based Decision Strategy | up to 24 weeks
  To calculate the Loss Frequency-Based Decision Strategy, a score will be calculated based on the preference for decks with low loss frequency (B + D) over decks with high loss frequency (A + C). A score greater than 0 indicates loss aversion, showing a preference for decks that present less frequent losses.
Learning | up to 24 weeks
  The choice scores [number of advantageous choices (deck C + D) minus the number of disadvantageous choices (deck A + B)] will be calculated for each block of 20 trials. The range of possible choice scores was from -100 to +100 for each block.

IPD SHARING:
Plan to Share IPD: Undecided
I will review any request and decide later.